CLINICAL TRIAL: NCT04185428
Title: Investigating Integrative Therapies for Symptom Management in Adults With Acute Leukemia Undergoing High-grade MDS Induction Chemotherapy
Brief Title: Investigating Integrative Therapies for Symptom Management in Adults With Acute Leukemia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The PIs left the institution.
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB201903226
Record Dates: First submitted 2019-12-02; First posted 2019-12-04 (Actual); Last update posted 2025-04-07 (Actual); Status verified 2025-04

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Intervention Model Description: In this feasibility pilot and qualitative interview mixed methods study, quantitative data will be used to describe the distribution of changes over time for anxiety, pain and other common symptoms among intervention and standard care groups as well as measures of feasibility and acceptability for the study design and methods.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care with integrative therapy (Experimental): For the intervention group, an initial interview will be conducted and the Patient-Reported Outcomes Measurement Information System (PROMIS) and Memorial Symptom Assessment Scale (MSAS) questionnaires will be administered at enrollment. Integrative Therapies will then begin offering two to four sessions weekly. At 7, 14, and 21 days (+-2 days) after the start of induction chemotherapy, the PROMIS and the MSAS questionnaires will be administered again along with an acceptability questionnaire. At 21 (+-2) days after the start of induction chemotherapy, a second interview will be conducted.
  Interventions: Behavioral: Integrative Therapy
- Standard of care only (No Intervention): For the standard care group, an initial interview will be conducted and the PROMIS and MSAS questionnaires will be administered at enrollment. At 7, 14, and 21 days (+-2 days) after the start of induction chemotherapy, the PROMIS and the MSAS questionnaires will be administered again. At 21 days (+-2 days) after the start of induction chemotherapy, a second interview will be conducted.

INTERVENTIONS:
Behavioral: Integrative Therapy — still meditation, meditative movement, relaxation techniques, and massage therapy
  Arms: Standard of care with integrative therapy

SUMMARY:
This pilot study will use a mixed methods approach to evaluate the feasibility and acceptability of Integrative Therapies, a bedside service offering mindfulness-based interventions (still meditation, meditative movement, relaxation techniques, and massage therapy) as non-pharmacologic treatment for symptom management in newly diagnosed adult Acute Myeloid Leukemia (AML) patients undergoing induction chemotherapy

DETAILED DESCRIPTION:
UF Health Integrative Therapies inpatient program offers mindfulness-based interventions consisting of still meditation, meditative movement, relaxation techniques, and massage therapy to patients at the bedside. This mixed methods feasibility pilot aims to move toward optimal use of the Integrative Therapies service amongst AML patients undergoing induction chemotherapy by: 1) examining the feasibility and acceptability of this intervention and describing the distribution of variables, 2) developing a greater understanding of patient experience, and 3) exploring facilitators and barriers to engagement with the service. The investigators intend to use the data collected from this study to inform a subsequent multi-site study with a larger sample size and adjustments depending on the results from this investigation.

The study team will also explore the acceptability to participation in Integrative Therapies bedside service by conducting a qualitative, phenomenological thematic analysis of patient interviews. The intent of a convergent design is to merge the analyses of the quantitative and qualitative data that are gathered during the implementation of Integrative Therapies bedside service.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to local area Bone Marrow Transplant Unit or Hematology/Oncology during the study period
* Diagnosed with acute leukemia
* Receiving high-grade MDS induction chemotherapy
* Within first 3 days of chemotherapy initiation
* Age > 18 years
* Able to speak/read English

Exclusion Criteria:

-Altered mental status or diminished level of consciousness as established by daily progress note documented by health care provider, nursing assessment, or at the discretion of the Integrative Therapies practitioner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2023-08-09 (Actual); Primary Completion 2025-03-04 (Actual); Study Completion 2025-03-04 (Actual)

PRIMARY OUTCOMES:
Feasibility of Integrative Therapy - proportion agreeing to participate | baseline through 3 weeks
  at least 50% electing to join the intervention
Feasibility of Integrative Therapy - proportion of participants who complete at least 5 sessions | baseline through 3 weeks
  a 70% completion rate (indicated by the completion of 5 or more sessions)
Acceptability of Integrative Therapy | baseline through 3 weeks
  Distribution of responses to acceptability with an acceptability benchmark of at least 75% of Integrative Therapy group members "rating the program as acceptable" via the acceptability questionnaire. Likert scoring 1-5, wit h on as very low and 5 being very high.

CONTACTS AND LOCATIONS:
Overall Officials: Nosha Farhadfar, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No